CLINICAL TRIAL: NCT01283815
Title: Laparoscopic Management of Periappendicular Abscess - Randomized Controlled Trial
Brief Title: Laparoscopic Management of Periappendicular Abscess
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Mentula, Surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUSOper193
Record Dates: First submitted 2011-01-20; First posted 2011-01-26 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Appendicitis; Abdominal Abscess
Keywords: Laparoscopy; Drainage; Appendectomy
MeSH Terms: conditions — Appendicitis; Abdominal Abscess | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative management (Active Comparator): Patients are treated with intravenous Cefuroxime 1,5 g x 3 per day plus Metronidazole 500 mg x 3 per day. If the abscess is at least 3 cm in diameter percutaneous ultrasound guided drainage is performed.
  Interventions: Procedure: Conservative management with percutaneous drainage
- Laparoscopic appendectomy (Experimental): Laparoscopic appendectomy and laparoscopic drainage of the abscess. If appendectomy is not possible due to technical difficulties only laparoscopic drainage is performed. Patients are treated with the same antimicrobial therapy as the control group
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy and laparoscopic drainage of the abscess. If appendectomy is not possible due to technical difficulties only laparoscopic drainage is performed. Patients are treated with the same antimicrobial therapy as the control group (intravenous Cefuroxime 1,5 g x 3 per day plus Metronidazole 500 mg x 3 per day).
  Arms: Laparoscopic appendectomy
Procedure: Conservative management with percutaneous drainage — Patients are treated with intravenous Cefuroxime 1,5 g x 3 per day plus Metronidazole 500 mg x 3 per day. If the abscess is at least 3 cm in diameter percutaneous ultrasound guided drainage is performed.
  Arms: Conservative management

SUMMARY:
According to retrospective studies the conservative management of periappendicular abscess is associated with decreased complication and re-operation rate compared with open appendectomy. Large abscesses require percutaneous drainage. Sometimes percutaneous drainage is not possible because of anatomical position of the abscess and surgical treatment is needed. The purpose of this study is evaluate whether laparoscopic appendectomy is suitable for the first-line treatment in patients with periappendicular abscess.

The hypothesis of the study is that laparoscopic management of periappendicular abscess is suitable for the first-line treatment and it does not increase time of hospitalization or complication rate compared with conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Periappendicular abscess at least 2 cm in size

Exclusion Criteria:

* Missing written informed consent
* Antimicrobial therapy lasted over 24 hours before randomization
* Attempt of drainage before randomization
* Age over 80 years or under 18 years old
* Pregnancy
* Allergy to either Cefuroxime or Metronidazole
* Severe chronic disease, that substantially increases the risk for operative mortality
* Previous major intra-abdominal surgery, that may have caused intra-abdominal adhesions
* Carrier of a resistant bacterial strain
* Being institutionalized or hospitalized for at least 2 weeks before randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time of hospitalization within the first 60 days after randomization | Day 60 after randomization

SECONDARY OUTCOMES:
Need of additional interventions | Within the first 60 days after randomization
  Interventions include percutaneous drainage and operations
Residual abscess | On day 7 after randomization
Attempted procedure not successfully performed | During the first 24 hours after randomization
  In the laparoscopy group appendectomy was not possible. In the conservative group planned percutaneous drainage was not possible.
The number of complications | Within 60 days from randomization
  Any complication occurring within 60 days from randomization. Both medical and surgical complications are included.
Number recurrent abscesses | Within 60 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Panu Mentula, M.D. Ph.D., Principal Investigator — Department of Gastrointestinal Surgery, Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Meilahti Hospital, Helsinki, Finland